CLINICAL TRIAL: NCT00447291
Title: Evaluation of the Safety and Efficacy of Omega-3 Fish Oil Dietary Supplementation in Biometric Measurement, Lipid Profile, Serum Markers for Inflammation, and Insulin Resistance in Overweight Children and Adolescents
Brief Title: Safety & Efficacy of Omega-3 Fish Oil in Overweight Children & Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Zone Labs, Inc discontinue utilizing their fish oil supplement and frozen foods
Sponsor: Children's Heart Center (Industry)
Collaborators: Zone Laboratories, Inc. (Industry)
Responsible Party: Gary A. Mayman/ Principal investigator, Children's Heart Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 06.02.001
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2006-09

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Fish Oil
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Supplement: Omega-3 Fish Oil
Behavioral: Multi-Disciplinary Nutrition & Exercise program

SUMMARY:
Children with an excess in body weight, increase the risk of obesity-related co-morbidities and cardiovascular diseases. Childhood obesity may be due to diets laden with fat and lack of physical activity. Omega-3 fish oil is a supplementation that may promote a greater reduction of pro-inflammatory mediators; combined with exercise and nutritional regimens it may also help improve glycemic, lipid markers, and body composition in overweight children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Between 8-18 years old
* BMI ≥95th percentile
* Patient & parent/guardian consent to participate
* Attendance of Risk Factor Reduction lifestyle modification program

Exclusion Criteria:

* Major surgical Procedure within 1 year
* Significant cardiovascular disease or other morbidity that preclude patients from following dietary regimen or exercising.
* Mentally Challenged
* Currently taking fish oil supplements, unless 1 month wash-out period is achieved.
* Diabetes

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To compare effects between Omega 3 fish oil and placebo | 3 months
  To compare the effect of Omega 3 fish oil dietary supplementation versus placebo on biometric measurement, lipid profile, serum markers for inflammation and insulin resistance in overweight children and adolescents undergoing treatment with a low-glycemic load diet and exercise.

SECONDARY OUTCOMES:
To compare effects between Omega 3 fish oil and placebo | 3 months
  To compare the changes in weekly physical activity, biometrics measurements and body mass index between overweight children and adolescents receiving Omega 3 fish oil supplementation versus placeb

CONTACTS AND LOCATIONS:
Overall Officials: Gary A. Mayman, MD, Principal Investigator — Children's Heart Center
Locations (1):
- Children's Heart Center, Las Vegas, Nevada, United States